CLINICAL TRIAL: NCT04517461
Title: Coagulation and Vitamin K in Head and Neck Microvascular Free Flap Surgery
Acronym: MVL-COAG
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00718
Record Dates: First submitted 2020-07-03; First posted 2020-08-18 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2022-04

CONDITIONS: Head and Neck Cancer; Intraoperative Complications; Coagulation Disorder, Blood; Vitamin K Deficiency; Thrombosis; Anticoagulants and Bleeding Disorders; Head and Neck Procedural Complication
MeSH Terms: conditions — Head and Neck Neoplasms; Intraoperative Complications; Blood Coagulation Disorders; Vitamin K Deficiency; Thrombosis; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood. Blood plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head and neck free flap surgery patients: Patients undergoing head and neck microvascular free flap surgery at Skåne University Hospital, Lund, Sweden.

SUMMARY:
For patients with large head and neck tumors the recommended treatment, in many cases, is a combination of extensive surgery and postoperative radiotherapy. The surgical procedure involves resection of the tumor and reconstruction with a so called microvascular free flap, i.e. tissue transferred from for instance the arm or leg to the resection site. Complications of this complex procedure include, but are not limited to, bleeding and blood cloths (thrombosis) in the transferred tissue (free flap), which can cause very serious complications including need for further surgery and loss of the flap.

Routine blood tests can measure parts of the system that regulates bleeding and the forming of blood clots, the so called coagulation system, but these tests don't cover the whole system. There are however more advanced instruments, such as ROTEM, rotational thromboelastometry, which provide a more global view of the hemostatic potential of whole blood. ROTEM is one of few more advanced assays that can be analyzed in emergency situations in major hospitals. Other more advanced coagulation assays are thrombin generation and measurements of specific coagulation factors, several of which are vitamin K dependent. Vitamin K is essential in the coagulation system and also involved in many other physiological processes. Deficiency of this vitamin is common, but not well studied in patients undergoing head an neck free flap surgery.

The investigators plan to study ROTEM and other above mentioned coagulation parameters in patients undergoing major head and neck surgery including microvascular free flap reconstruction to assess if these parameters can help predict patients at risk for bleeding or flap thrombosis. Further on this could hopefully enable prevention of complications and improve treatment of coagulation complications that still occur.

DETAILED DESCRIPTION:
Microvascular reconstructive free flap surgery is an important part of the recommended treatment for extensive head and neck tumors. However, the procedure includes risks of perioperative coagulation related complications, such as bleeding, but also thrombosis in the flap blood vessels. In about 10% of cases this requires reoperation, but, in spite of intense efforts, about 5% of all patients suffer from flap failure, i.e. necrosis of the free flap. This results in significant suffering for the patients who must undergo further surgery and oftentimes considerable prolonged hospital stay etc. This in turn leads to increased health care costs. There are several indications that tendency towards thrombosis can increase the risk of flap failure.

Previous studies have indicated that increased levels of fibrinogen and inherited thrombophilia, such as APC resistance, are associated with thrombotic free flap complications, but more conventional coagulation parameters, such as PK/INR and aPTT have not shown the same connection. Low fibrinogen levels have also been associated with bleeding complications.

Most patients undergoing the above mentioned surgery receive anticoagulant therapy. However, there is no international consensus on any specific pharmacological regime. Many different prophylactic therapies are used, including low molecular weight heparin, dextran and acetylsalicylic acid. Still coagulation-related complications are difficult to prevent.

Defective coagulation apparently seems to be associated with bleeding and thrombotic perioperative complications. It would therefore be desirable to increase the knowledge about factors influencing the development of these complications, and the patients at risk for them. ROTEM, rotational thromboelastometry, is a viscoelastic essay that provides a more global view of the hemostatic potential in whole blood, and it is also one of few more advanced assays that can be analyzed around the clock in many Swedish hospitals.

The aim of this project is to study perioperative coagulation and vitamin K status, and thereby further on hopefully be able to prevent, and improve the treatment of, bleeding and thrombosis related complications in patients undergoing head and neck microvascular free flap surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing head and neck surgery including resection and reconstruction with a microvascular free flap at Skåne University Hospital in Lund, Sweden, who accept participation in the study.

Exclusion Criteria:

* Age under 18 years.
* Inability to understand information or make an informed choice about participation.
* Hospitalization > 24 h prior to primary surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that present at, or are referred to, the Department of Otorhinolaryngology - Head and Neck Surgery at Skåne University Hospital in Lund with conditions requiring head and neck surgery including resection and reconstruction with a microvascular free flap. This includes patients from the entire southern health care region, "Södra sjukvårdsregionen".
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Perioperative changes in ROTEM MCF EXTEM | Day 0 to day 6
  Perioperative changes in ROTEM MCF (EXTEM). Baseline values measured at start of surgery (day 0), thereafter repeated measurements are made until day 6. Power calculation is based on an expected change in ROTEM MCF (EXTEM) from day 0 to postoperative day 2 (based on Lison et al, Blood Coagul Fibrinolysis. 2011.).

SECONDARY OUTCOMES:
Perioperative changes in ROTEM Clotting time | Day 0 to day 6
  Perioperative changes in ROTEM Clotting Time (CT, s). Baseline values measured at start of surgery (day 0), thereafter repeated measurements are made until day 6.
Perioperative changes in ROTEM Clot Formation Time | Day 0 to day 6
  Perioperative changes in ROTEM Clot Formation Time (CFT, s).
Perioperative changes in ROTEM alpha angle | Day 0 to day 6
  Perioperative changes in ROTEM alpha angle (°).
Perioperative changes in ROTEM Lysis Index 60 | Day 0 to day 6
  Perioperative changes in ROTEM Lysis Index 60 (LI60, %).
Perioperative changes in ROTEM Maximum Clot Firmness | Day 0 to day 6
  Perioperative changes in ROTEM Maximum Clot Firmness (mm).
Perioperative changes in prothrombin time | Day 0 to day 6
  Perioperative changes in prothrombin time (INR).
Perioperative changes in activated partial thromboplastin time | Day 0 to day 6
  Perioperative changes in activated partial thromboplastin time (APTT, s).
Perioperative changes in thrombocyte levels | Day 0 to day 6
  Perioperative changes in thrombocyte levels (number/L).
Perioperative changes in thrombin generation; lag time | Day 0 to day 6
  Perioperative changes in thrombin generation; lag time (s).
Perioperative changes in thrombin generation; peak thrombin | Day 0 to day 6
  Perioperative changes in thrombin generation; peak thrombin (nM).
Perioperative changes in thrombin generation; area under the curve | Day 0 to day 6
  Perioperative changes in thrombin generation; area under the curve (AUC).
Perioperative changes in specific coagulation factors; protein C (kIU/L) | Day 0 to day 6
  Perioperative changes in protein C (kIU/L).
Perioperative changes in specific coagulation factors; protein S | Day 0 to day 6
  Perioperative changes in protein S (kIU/L).
Perioperative changes in specific coagulation factors; fibrinogen | Day 0 to day 6
  Perioperative changes in fibrinogen (g/L).
Perioperative changes in specific coagulation factors; antithrombin | Day 0 to day 6
  Perioperative changes in antithrombin (kIU/L).
Perioperative changes in fibrinolytic activation | Day 0 to day 6
  Perioperative changes in plasmin-antiplasmin complex, PAP (μg/L).
Perioperative changes in the vitamin K-dependent protein Gas6 | Day 0 to day 6
  Perioperative changes in the vitamin K-dependent protein Gas6 (ng/mL).
Perioperative changes in the vitamin K-dependent protein dp-uc-MGP | Day 0 to day 6
  Perioperative changes in the vitamin K-dependent protein dp-uc-MGP (pM/L).
Perioperative changes in the vitamin K-dependent protein Axl-receptor | Day 0 to day 6
  Perioperative changes in the vitamin K-dependent protein Axl-receptor (pg/mL).
Perioperative changes in the vitamin K-dependent protein PIVKA-II | Day 0 to day 6
  Perioperative changes in the vitamin K-dependent protein PIVKA-II (mAU/mL).
Coagulation related complications | Day 0 until end of hospital stay or a at the latest day 30 days after the primary operation.
  Connection between perioperative complications (thrombotic [arterial/venous] or bleeding) in the surgical site and abnormal levels of coagulation parameters mentioned above.
Perioperative changes in ROTEM FIBTEM Maximum Clot Firmness | Day 0 to day 6
  Perioperative changes in ROTEM INTEM Maximum Clot Firmness (MCF, mm).
Perioperative changes in ROTEM INTEM Clotting Time | Day 0 to day 6
  Perioperative changes in ROTEM INTEM Clotting Time (CT, s).

CONTACTS AND LOCATIONS:
Overall Officials: Caroline U Nilsson, MD, PhD, Study Chair — Skane University Hospital
Locations (1):
- Region Skåne, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cervenka B, Bewley AF. Free flap monitoring: a review of the recent literature. Curr Opin Otolaryngol Head Neck Surg. 2015 Oct;23(5):393-8. doi: 10.1097/MOO.0000000000000189. PMID 26339970
- [Background] Copelli C, Tewfik K, Cassano L, Pederneschi N, Catanzaro S, Manfuso A, Cocchi R. Management of free flap failure in head and neck surgery. Acta Otorhinolaryngol Ital. 2017 Oct;37(5):387-392. doi: 10.14639/0392-100X-1376. PMID 29165433
- [Background] Kolbenschlag J, Daigeler A, Lauer S, Wittenberg G, Fischer S, Kapalschinski N, Lehnhardt M, Goertz O. Can rotational thromboelastometry predict thrombotic complications in reconstructive microsurgery? Microsurgery. 2014 May;34(4):253-60. doi: 10.1002/micr.22199. Epub 2013 Oct 21. PMID 24142816
- [Background] Lison S, Weiss G, Spannagl M, Heindl B. Postoperative changes in procoagulant factors after major surgery. Blood Coagul Fibrinolysis. 2011 Apr;22(3):190-6. doi: 10.1097/MBC.0b013e328343f7be. PMID 21245747
- [Background] Handschel J, Burghardt S, Naujoks C, Kubler NR, Giers G. Parameters predicting complications in flap surgery. Oral Surg Oral Med Oral Pathol Oral Radiol. 2013 May;115(5):589-94. doi: 10.1016/j.oooo.2012.09.007. Epub 2012 Dec 12. PMID 23246227
- [Background] Kolbenschlag J, Diehm Y, Daigeler A, Kampa D, Fischer S, Kapalschinski N, Goertz O, Lehnhardt M. Insufficient fibrinogen response following free flap surgery is associated with bleeding complications. GMS Interdiscip Plast Reconstr Surg DGPW. 2016 Nov 22;5:Doc22. doi: 10.3205/iprs000101. eCollection 2016. PMID 27975041
- [Background] Zhou W, Zhang WB, Yu Y, Wang Y, Mao C, Guo CB, Yu GY, Peng X. Are antithrombotic agents necessary for head and neck microvascular surgery? Int J Oral Maxillofac Surg. 2019 Jul;48(7):869-874. doi: 10.1016/j.ijom.2018.10.022. Epub 2018 Nov 26. PMID 30497789